CLINICAL TRIAL: NCT05777759
Title: A Randomized, Evaluator-blinded, Parallel Group, Comparator-controlled, Multicenter Study to Evaluate the Safety and Effectiveness of Restylane Lyft With Lidocaine for Augmentation of the Chin Region to Improve the Chin Profile
Brief Title: Safety and Effectiveness of Restylane Lyft With Lidocaine for Augmentation of the Chin Region to Improve the Chin Profile
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43USCH2208
Record Dates: First submitted 2023-03-09; First posted 2023-03-21 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Chin Augmentation; Chin Retrusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- New Dermal Filler for indication: Restylane Lyft with Lidocaine (Experimental): hyaluronic acid dermal filler
  Interventions: Device: Restylane Lyft with Lidocaine
- Active Comparator: FDA approved Dermal Filler: Juvederm Voluma XC (Active Comparator): hyaluronic acid dermal filler
  Interventions: Device: Juvederm Voluma XC

INTERVENTIONS:
Device: Restylane Lyft with Lidocaine — hyaluronic acid
  Arms: New Dermal Filler for indication: Restylane Lyft with Lidocaine
Device: Juvederm Voluma XC — hyaluronic acid
  Arms: Active Comparator: FDA approved Dermal Filler: Juvederm Voluma XC

SUMMARY:
The primary objective of the study is to demonstrate non-inferiority of Restylane Lyft with Lidocaine versus a comparator-control for augmentation of the chin region to improve the chin profile.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant, non-breastfeeding females, 22 years of age or older
* Intent to receive treatment for augmentation and correction of retrusion in the chin region.

Exclusion Criteria:

* Known/previous allergy of hypersensitivity to any injectable hyaluronic acid (HA) gel or gram-positive bacterial proteins.
* Known/previous allergy or hypersensitivity to local anesthetics, e.g., lidocaine or other amide-type anesthetics.
* Previous or present multiple severe allergies or severe allergies, such as manifested by anaphylaxis or angioedema or family history of angioedema.
* Previous facial surgery (including facial aesthetic surgery and liposuction), below the level of the horizontal line from the subnasale.
* Any previous aesthetic procedures or implants
* Presence of any disease or lesion near or on the area to be treated.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-11-11 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Primary Effectiveness Objective | 3 months after last treatment
  Change from Baseline in the Blinded Evaluators' live assessment using the GCRS (Galderma Chin Retrusion Scale).

SECONDARY OUTCOMES:
Secondary Effectiveness Objective | 6, 9, and 12 months after last treatment.
  Responder rate based on the Blinded Evaluator's live assessment using the GCRS (Galderma Chin Retrusion Scale) at 6, 9, and 12 months after last treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (12):
- United States (11):
  - Galderma Research Site, Los Angeles, California
  - United States, California, Manhattan Beach, California
  - Galderma Research Site, Westport, Connecticut
  - Galderma Research Site, Aventura, Florida
  - Galderma Research Site, Coral Gables, Florida
  - Galderma Research Site, Alpharetta, Georgia
  - Galderma Research Site, Atlanta, Georgia
  - Galderma Research Site, Rockville, Maryland
  - Galderma Research Site, Chestnut Hill, Massachusetts
  - Galderma Research Site, Nashville, Tennessee
  - Galderma Research Site, Pflugerville, Texas
- Galderma Research Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No